CLINICAL TRIAL: NCT05298332
Title: A Phase 1, Open-Label, 3-Cohort, Parallel, Single Dose Study of the Safety, Tolerability, and Pharmacokinetics of a Single Oral Dose ATI-2173 50 mg in Healthy Japanese, Chinese, and Non-Asian Subjects
Brief Title: Ethnobridging Study in Healthy Volunteers, Chinese and Japanese Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated by the Sponsor
Sponsor: Antios Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANTT104
Record Dates: First submitted 2022-02-24; First posted 2022-03-28 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ATI-2173 50 mg Japanese (Experimental): Healthy adult Japanese subjects will receive 50 mg of ATI-2173
  Interventions: Drug: ATI-2173 50 mg
- ATI-2173 50 mg Chinese (Experimental): Healthy adult Chinese subjects will receive 50 mg of ATI-2173
  Interventions: Drug: ATI-2173 50 mg
- ATI-2173 50 mg Non-Asian (Experimental): Healthy adult non-Asian subjects will receive 50 mg of ATI-2173
  Interventions: Drug: ATI-2173 50 mg

INTERVENTIONS:
Drug: ATI-2173 50 mg — ATI-2173 is a phosphoramidate prodrug of the oral, non-chain terminating nucleoside analog clevudine being developed by Antios Therapeutics, Inc. for treatment of men and women with chronic hepatitis B (CHB)

SUMMARY:
This is a single center, open-label, 3-Cohort, parallel, single-dose, study to evaluate the PK, safety, and tolerability of ATI-2173 50 mg administered orally in Japanese, Chinese, and Non-Asian healthy subjects incorporating a food effect analysis in Non-Asian healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures (including ability and willingness to abstain from alcohol from 48 hours prior to the first study drug administration until discharge) and availability for the duration of the study
3. Healthy adult male or female
4. Aged between 18 and 59 years, inclusive
5. Weight ≥ 50.0 kg and ≤ 100 kg
6. Body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively
7. Non- or ex-smoker (an ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration)
8. Suitable veins for cannulation or repeated venipuncture as assessed by an Investigator at Screening
9. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an Investigator
10. Agrees to abstain from blood or plasma donation from the Screening visit until 3 months after the last study drug administration
11. If female, must meet one of the following criteria:

    1. Is of childbearing potential and agrees to use an acceptable contraceptive method.

       Acceptable contraceptive methods include:
       * Abstinence from heterosexual intercourse from Screening through to at least 60 days after the last study drug administration
       * Male partner vasectomized at least 180 days prior to Screening
       * Double-barrier method (eg, male condom, spermicide and diaphragm or male condom, spermicide and cervical cap used simultaneously) from Screening through to at least 30 days after the last study drug administration
       * One of the following contraceptive methods with a barrier method (eg, male condom) from at least 28 days prior to the first study drug administration through to at least 60 days after the last study drug administration:
       * Systemic contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
       * Intrauterine device (with or without hormones) OR
    2. Is of non-childbearing potential, defined as surgically sterile (ie, has undergone complete hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or tubal ligation/occlusion) or in a postmenopausal state (at least 1 year without menses without an alternative medical condition prior to Screening), as confirmed by follicle-stimulating hormone levels (≥ 40 mIU/mL).
12. A male study subject that engages in sexual activity that has the risk of pregnancy must:

    * Agree to use a double-barrier method (eg, male condom, spermicide, and diaphragm or male condom, spermicide, and cervical cap used simultaneously) if female partner is of child-bearing potential or be abstinent from heterosexual intercourse from Screening to at least 90 days after the last study drug administration or be unable to procreate; defined as surgically sterile (i.e. has undergone a vasectomy at least 180 days prior to Screening AND
    * Agree to not donate sperm during the study and for at least 90 days after the last study drug administration.

    For Cohort 1 only:
13. The subject must have been born in Japan and have both parents and 4 grandparents of Japanese descent.
14. The subject must have lived outside of Japan for no more than 10 years.
15. The subject must have not significantly changed their diet and lifestyle since leaving Japan.

    For Cohort 2 only:
16. The subject must have been born in China or Chinese subjects who were born in Taiwan, Hong Kong, Macau, Mongolia, or Singapore and have both parents and 4 grandparents of Chinese descent.
17. The subject must have lived outside of Chinese for no more than 10 years.
18. The subject must have not significantly changed their diet and lifestyle since leaving China.

    For Cohort 3 only:
19. The subjects must be of Non-Asian descent, as evidenced by verbal confirmation that both parents and all 4 grandparents are Non-Asian.

Exclusion Criteria:

1. Female who is lactating
2. Female who is pregnant according to the pregnancy test at Screening or prior to the first study drug administration
3. Blood pressure and pulse rate outside normal range and clinically significant at Screening or prior to the first study drug administration, in the opinion of an Investigator
4. History of hypersensitivity to ATI-2173 or clevudine, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
5. Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability including but not limited to cholecystectomy (excluding appendectomy)
6. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease, in the opinion of an Investigator
7. Presence of clinically significant ECG abnormalities at Screening or prior to the first study drug administration, in the opinion of an Investigator
8. Presence of clinically significant muscle disorders, myopathies or other forms of liver disease, in the opinion of an Investigator
9. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 using the Modification of Diet in Renal Disease (MDRD) equation at Screening or prior to the first study drug administration
10. Unexplained persistent elevations of serum transaminases or creatine kinase (CK) levels that are clinically significant per Investigator discretion, at Screening or prior to the first study drug administration
11. Immunization with a Coronavirus Disease 2019 (COVID-19) vaccine in the 14 days prior to the first study drug administration
12. Scheduled immunization with a COVID-19 vaccine (first, second or booster dose) during the study that, in the opinion of an Investigator, could potentially interfere with subject participation, subject safety, study results, or any other reason
13. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
14. Any clinically significant illness in the 28 days prior to the first study drug administration
15. Use of any prescription drugs (except systemic contraception and intrauterine devices), including but not limited to inducers, inhibitors, or substrates of P-glycoprotein and CYP3A4, in the 28 days prior to the first study drug administration, that in the opinion of an Investigator would put into question the status of the participant as healthy or that could potentially interact with the study drug
16. Use of St. John's wort in the 28 days prior to the first study drug administration
17. Any history of tuberculosis
18. Use of quinine-containing products (eg, tonic water), grapefruit products, pomelo products, Seville orange products, including supplements containing Citrus aurantium or "bitter orange", in the 14 days prior to the first study drug administration
19. Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first study drug administration
20. Positive test results for HIV-1/HIV-2 antibodies, hepatitis B surface antigen or hepatitis C antibody at Screening
21. Any other clinically significant abnormalities in laboratory test results at Screening or prior to the first study drug administration that would, in the opinion of an Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
22. Inclusion in a previous group for this clinical study
23. Participation in another clinical study with a non-biologic Investigational Product (IP) or new formulation of a marketed non-biologic drug in the 30 days prior to dosing
24. Participation in another clinical study with a biologic (marketed or investigational) in the 90 days or 5 half-lives (whichever is longer) prior to dosing
25. Donation of plasma in the 7 days prior to Screening
26. Donation of 1 unit of blood to American Red Cross or equivalent organization or donation of over 500 mL of blood in the 56 days prior Screening

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Cmax of ATI-2173, clevudine, and M1 in plasma | Through the end of study, average of 3 months
Tmax ATI-2173, clevudine, and M1 in plasma | Through the end of study, average of 3 months
AUC0-t ATI-2173, clevudine, and M1 in plasma | Through the end of study, average of 3 months
AUC0-inf ATI-2173, clevudine, and M1 in plasma | Through the end of study, average of 3 months
T1/2 ATI-2173, clevudine, and M1 in plasma | Through the end of study, average of 3 months
CL/F of ATI-2173, clevudine, and M1 in plasma | Through the end of study, average of 3 months
Vz/F of ATI-2173, clevudine, and M1 in plasma | Through the end of study, average of 3 months
Ae of ATI-2173, clevudine, and M1 in urine | Through the end of study, average of 3 months
CLR of ATI-2173 in urine | Through the end of study, average of 3 months
mCLR of clevudine, and M1 in urine | Through the end of study, average of 3 months

SECONDARY OUTCOMES:
Number of adverse events | Through the end of study, average of 3 months
Cmax of ATI-2173, clevudine, and M1 in plasma for food effect | Through the end of study, average of 3 months
AUC0-72 of ATI-2173, clevudine, and M1 in plasma for food effect | Through the end of study, average of 3 months
AUC0-inf of ATI-2173, clevudine, and M1 in plasma for food effect | Through the end of study, average of 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences, Cypress, California, United States